CLINICAL TRIAL: NCT07029256
Title: Ultrasound-Guided Core Needle Biopsy to Stage Urothelial Carcinoma of the Bladder
Brief Title: Ultrasound-Guided Core Needle Biopsy to Stage Urothelial Carcinoma of the Bladder (US UCB)
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 23-008092; NCI-2024-09054 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23-008092 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2025-06-10; First posted 2025-06-19 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Bladder Urothelial Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Bladder tissue

GROUPS / COHORTS (1):
- Observational: Patients undergo standard of care radical cystectomy and residual tissues collected undergo US core needle biopsy. Additionally, patients have their medical records reviewed on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study is being done to test the feasibility and accuracy of using an ultrasound-guided core needle biopsy technique as a potential tool for staging urothelial carcinoma of the bladder (UCB).

ELIGIBILITY:
Inclusion Criteria:

* Undergoing radical cystectomy for confirmed or suspected urothelial carcinoma of the bladder
* Prior abdominal imaging

Exclusion Criteria:

* History of partial cystectomy or complex bladder reconstruction or substitution (i.e. bladder augment or urothelial recurrence in a neobladder)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing radical cystectomy for confirmed or suspected urothelial carcinoma of the bladder
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-26 (Actual); Primary Completion 2030-07-30 (Estimated); Study Completion 2030-07-30 (Estimated)

PRIMARY OUTCOMES:
Concordance between US and core needle biopsy stage and final surgical specimen pathologic stage | Baseline (after completion of bladder surgery)
  The radiology-assessed tumor stage from the ultrasound (US) and the core needle biopsy-assessed tumor stage will be compared with the final pathologic tumor stage.

CONTACTS AND LOCATIONS:
Overall Officials: Vidit Sharma, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials